CLINICAL TRIAL: NCT06372951
Title: Role of Lung Ultrasound in Assessment of Neonatal Respiratory Distress
Brief Title: Lung Ultrasound in Neonatal Intensive Care Units
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Talat Fawzy, : Assistant Lecturer, Assiut University
Other Study IDs: Lung ultrasound in neonate
Record Dates: First submitted 2023-11-29; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Neonatal Respiratory Distress
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound — A device that use ultrasonic waves as a way to image the internal organs and tissues of the body in order to diagnose the different diseases.

SUMMARY:
Identification of lung diseases causing neonatal respiratory distress by lung ultrasound as a tool that can replace x-ray .

DETAILED DESCRIPTION:
* Lung disease is the most common cause of neonatal respiratory distress.
* It can result in respiratory failure and death in severe cases.
* The mortality rate is approximately 11%:32%.
* Identification of the etiology of lung disease is important for neonatologists.
* Traditionally, chest X-ray has been considered as the most valuable imaging modality for the diagnosis of lung diseases, but it unavoidably causes radiation damage to the patient.
* Neonates are susceptible to radiation because they have rapidly dividing cells that cannot repair mutated DNA.
* The risk of cancer induction in infants receiving a single small dose of radiation is 2-3 times higher than the average population and 6-9 times higher than the risk from an exposure of a 60-year-old patient.
* New imaging modalities have been introduced in clinical practice in recent years such as lung ultrasound.
* One of the most common causes of neonatal respiratory distress that can be diagnosed by ultrasound is :Respiratory Distress Syndrome:

  * Respiratory distress syndrome.. is a major cause of neonatal mortality.
  * It mainly occur in preterm infants due to structural and functional lung immaturity.
  * Pulmonary surfactant insufficiency is an important pathogenesis in respiratory distress syndrome.
  * The ultrasonic features of respiratory distress syndrome are: Compact B-Lines, white lung appearance, abnormality in pleural line (thick and irregular),lung consolidation.
* Lung ultrasound has the advantages of :

  * Non-ionizing.
  * Easy to operate.
  * Low coast.
  * Portable for bedside use.
  * The imaging is performed in real-time.
* Thus making it as a potential tool to be used in neonatal intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* Neonates in neonatal intensive care units

Exclusion Criteria:

* Patients with poor-quality of lung ultrasound image.
* Subcutaneous emphysema.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Nenates in the neonatal intensive care units who suffering from respiratory distress.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Identifying causes of neonatal respiratory distress | Baseline
  - To evaluate lung ultrasound accuracy and reliability in diagnosing pulmonary disease in neonates in comparison to x rays

CONTACTS AND LOCATIONS:
Overall Officials: Ihab Mansour Mohamed, Prof., Study Director — Assiut University; Kawsar Abdel Halim Mohamed, Lecturer, Study Director — Assiut University; Azhar Arabi Mohammed, Lecturer, Study Director — Assiut University